CLINICAL TRIAL: NCT05207553
Title: Validity and Test Re-test Reliability of the Urdu Version of Lysholm Knee Scoring Scale in Patients With Anterior Cruciate Ligament Injuries in the Pakistani Clinical Setting.
Brief Title: A Reliability and Validity Study of Urdu Version of Lysholm Knee Scoring Scale.
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0286
Record Dates: First submitted 2022-01-24; First posted 2022-01-26 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Lysholm Knee Scale; Anterior Cruciate Ligament Injuries; Knee disorders; Validity; Urdu Version; Reliability; Arthroscopic Knee
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will be intended to translate and check if the Urdu Version of Lysholm Knee Scoring Scale is reliable and valid in the Pakistani patients with anterior cruciate ligament injuries.

DETAILED DESCRIPTION:
A detailed research will be conducted on nearly 100 patients after ethical approval from the Ethical Review Board of Riphah International University Faisalabad Campus. A total of 100 patients with Anterior Cruciate Ligament injuries will be selected from different areas of community and rehabilitation centers. Informed consent will be taken from each patient. The tool will be used three times in the same Pakistani population with Anterior Cruciate Ligament injuries to check inter and intra-observer reliability of the final Urdu-LKS. The Lysholm questionnaire translation will be carried out in 6 steps by the guidelines of the early researches and the Consensus-based Standards for the selection of health Measurement Instruments standard. Statistical Package of Social Sciences 23 will be employed to do data analysis.

ELIGIBILITY:
Inclusion Criteria:

* From17 years Old to 60 Years Old
* Presence of an Anterior Cruciate Ligament Injury or Ligament Repair
* No intervention between the test-retest assessments.

Exclusion Criteria:

* To complete the forms because of a psychological Impairment.
* Illiteracy or lack of understanding of Urdu Language
* Had a condition that couldn't be settled after a second assessment for different sicknesses like cancer, any other serious Infection, or inflammatory disease
* The presence of neurologic or musculoskeletal disorders other than the knee Condition.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pakistani population with anterior cruciate ligament injuries was included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Lysholm Knee Scoring Scale | 1st day
  • The Lysholm scale was developed for use by physicians and has been verified in patients with Anterior Cruciate Ligament and meniscal injuries. It's also been approved as a patient-administered tool for assessing symptoms and function in people who have had a variety of knee injuries. The Lysholm scale assesses the domains of symptoms and complaints, as well as functioning in daily activities, however, it doesn't assess the area of sports and recreational activities. There are 8 items on this questionnaire and graded on a scale of 0 to 100, with higher scores suggesting fewer symptoms and better function.
Kujala Anterior Knee Pain Scale | 1st day
  Kujala Anterior Knee Pain Scale - a patient-reported evaluation of subjective symptoms and functional limitations in patients with patellofemoral diseases, was published. Patients with anterior knee pain, patellar subluxation, and patellar dislocation, as well as a control group, were included in the initial study group for the score. The Kujala questionnaire has 13 items totaling 100 points. All 13 questions in the original 1993 study had statistically significant between-group differences.
International Knee Documentation Committee Questionnaire | 1st day
  The IKDC is a patient-completed questionnaire that comprises sections on tibiofemoral joint physical signs (7 items), function (2 items), and sports activities (3 things) (2 items). Scores vary from 0 to 100, with 0 being the lowest degree of function and 100 demonstrating the uppermost level of physical signs.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No